CLINICAL TRIAL: NCT05452226
Title: Neuromuscular Electrical Stimulation (NMES) in Patients Hospitalized With Acute Exacerbation of COPD and/or Community Acquired Pneumonia
Brief Title: Neuromuscular Electrical Stimulation in COPD/Community Acquired Pneumonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Renee Stapleton, Professor of Medicine, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002023
Record Dates: First submitted 2022-06-14; First posted 2022-07-11 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-02

CONDITIONS: Community-acquired Pneumonia; COPD Exacerbation Acute
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Intervention Model Description: small, prospective cohort study where every participant receives the study intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Pilot Study Cohort (Experimental): Every participant in this small prospective cohort study will receive the study intervention.
  Interventions: Device: neuromuscular electrical stimulation (NMES)

INTERVENTIONS:
Device: neuromuscular electrical stimulation (NMES) — Electrical stimulation will be applied using two adhesive pads affixed to the front of both of the thighs. The intensity will be progressively increased to a level that provokes a strong contraction. The stimulation intensity will be increased until the stimulation is uncomfortable, but does not hurt. Care will be taken to make sure that the level of stimulation will be adjusted such that the intensity does not cause pain. Contractions will last 10 seconds, with 30 seconds of rest between. NMES will occur 6 days per week for 60 minutes per day. Patients will self-administer NMES 6 days per week after discharge for up to 6 weeks.

SUMMARY:
In older adults hospitalized for acute medical conditions, immobility, clinical treatments, and the illness itself contribute to physical deconditioning and delirium, hospital-acquired impairments that increase risk for long-term physical and mental disability, other morbidities, and death. In patients with acute respiratory failure, hospital-acquired functional impairments persist long after hospitalization, due to limited use to rehabilitative interventions in the inpatient or post-acute settings. Exercise and early mobilization interventions are safe and improve physical and cognitive impairments, but there are critical barriers to their widespread implementation in acute care and home settings, including mobility limitations, reduced cardiopulmonary reserve, limited staff, and costs. Thus, there is an unmet need to develop interventions that can be utilized in both the inpatient and home environments to improve functional recovery in patients with acute exacerbation of chronic obstructive pulmonary disease (AECOPD) and community-acquired pneumonia (CAP).

This study addresses this clinical need and these barriers and will provide important feasibility and acceptability data regarding the utility of neuromuscular electrical stimulation (NMES) administered to lower extremity musculature across inpatient and post-discharge settings to improve functional and cognitive recovery in older adults hospitalized for AECOPD/CAP.

Initial NMES sessions will begin during participants' stay at UVM Medical Center and will continue at home after hospital discharge. Study participants will be issued a portable NMES device to take home and instructed on its use. They will receive guidance and oversight on the use of the NMES device and will be asked to perform NMES treatments 6 days per week for 60 minutes per day for 6 weeks. Data will be collected via activity monitor, participant questionnaires and clinical assessments including strength testing and 6-minute-walk-test.

DETAILED DESCRIPTION:
In older adults hospitalized for acute medical conditions, immobility, clinical treatments, and the illness itself contribute to physical deconditioning and delirium, hospital-acquired impairments that increase risk for long-term physical and mental disability, other morbidities, and death1-11. The syndrome of "long COVID" has drawn attention to the physical and psychological sequelae of hospitalization for acute respiratory illness (ARI), but this is not a new phenomenon. In patients with ARI, hospital-acquired functional impairments persist long after hospitalization, due to limited use to rehabilitative interventions in the inpatient or post-acute settings12-14. Exercise and early mobilization interventions are safe15 and improve physical and cognitive impairments16-19, but there are critical barriers to their widespread implementation in acute care and home settings, including mobility limitations, reduced cardiopulmonary reserve, limited staff, and costs. Thus, novel, interventions are needed that are portable, easy to use, and require minimal costs and equipment.

Community-acquired pneumonia (CAP) and acute exacerbation of chronic obstructive pulmonary disease (AECOPD) are leading causes of hospitalization in older adults20. These diagnoses often overlap21, cause substantial morbidity and mortality, and together account for >2.5 million hospitalizations and >$80 billion in costs annually22-28. Even before the COVID global pandemic, disability after hospitalization for AECOPD/CAP was on the rise29, due, in part, to an inability to remediate hospital-acquired impairments secondary to the lack of availability and low utilization of rehabilitation interventions13,30.

Physical rehabilitation improves mobility and attenuates hospital-acquired disability16-18, but these services are limited and their utilization in the hospital and after discharge is low. For instance, rehabilitation programs are absent or grossly underutilized for most general medical conditions, such as CAP. Even among patients with COPD, where rehabilitation has well-proven benefits and is supported by third party payers, uptake of pulmonary rehabilitation (PR) after hospitalization is very poor, with <3% participation within 1 year13. Low utilization of these services is due, in part, to barriers to delivering rehabilitation interventions in patient populations in the acute and post-discharge care settings, including inadequate staffing, costs, disease symptoms, reduced cardiopulmonary reserve, and lack of facility-based programs. Thus, there is an unmet need to develop interventions that can be utilized in both the inpatient and home environments to improve functional recovery in patients with AECOPD/CAP.

This study addresses this clinical need and these barriers and will provide important feasibility and acceptability data regarding the utility of neuromuscular electrical stimulation (NMES) administered to lower extremity musculature across inpatient and post-discharge settings to improve functional and cognitive recovery in older adults hospitalized for AECOPD/CAP.

ELIGIBILITY:
Inclusion Criteria:

1. >50 years old
2. Hospitalized for CAP and/or AECOPD
3. Expected hospital stay >2 days after enrollment (to permit adequate application of and training in NMES)

Exclusion Criteria:

1. >7 days of hospitalization prior to enrollment
2. Life expectancy < 6 months
3. Clinical Frailty Scale87 score >6
4. Lower extremity impairments that prevent bilateral use of NMES (e.g., amputation, leg injury)
5. Acute lower extremity deep vein thrombosis
6. Implanted cardioverter-defibrillator or pacemaker
7. Body mass index (BMI) >40 kg/m2
8. Currently requiring ICU care (including for sepsis)90. Prior ICU care during this hospitalization acceptable.
9. Severe skin breakdown on either lower extremity
10. Not ambulating independently prior to admission (gait aid is permitted)
11. New or existing intracranial, spinal, vascular, or neuromuscular condition limiting walking ability
12. Language barrier prohibiting outcome assessment
13. More than mild pre-existing dementia (IQCODE* score >3.6)
14. Likely discharge to setting where study team cannot oversee/monitor intervention (e.g., skilled nursing facility where team cannot monitor compliance)
15. Incarcerated
16. Refuses informed consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility assessed by study recruitment | 6 weeks
  recruitment of n=8 patients
Feasibility assessed by outcome assessment completion | 6 weeks
  completion of ≥90% of secondary outcome assessments
Feasibility assessed by adherence to the intervention | 6 weeks
  adherence to NMES of ≥80% during hospitalization and ≥60% at home
Acceptability as assessed by a NMES-specific questionnaire | 6 weeks
  Acceptability of the NMES intervention will be measured using a 10-item questionnaire that uses a Likert rating scale developed by our group for use with NMES, with 5 items allowing further qualitative input from volunteers to identify action items for improving delivery of the NMES intervention.

SECONDARY OUTCOMES:
physical functioning: ability to walk independently | enrollment, time of hospital discharge up to 6 weeks, 6 week follow-up
  6 minute walk test (6MWT)
physical functioning: mobility of the lower extremity | enrollment, time of hospital discharge up to 6 weeks, 6 week follow-up
  short physical performance battery (SPPB)
knee extensor torque | enrollment, time of hospital discharge up to 6 weeks, 6 week follow-up
  isometric dynamometry

CONTACTS AND LOCATIONS:
Overall Officials: Renee Stapleton, MD, PhD, Principal Investigator — University of Vermont Department of Medicine
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No